CLINICAL TRIAL: NCT05631496
Title: Validity and Reliability of the Turkish Marx Activity Rating Scale for Knee Disorders
Brief Title: Validity and Reliability of Turkish Version of Marx Activity Rating Scale
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Other Study IDs: Yeditepe U
Record Dates: First submitted 2022-11-21; First posted 2022-11-30 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-01

CONDITIONS: Knee Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with Knee Disorders: Patients with knee disorders such as traumatic meniscal and ligament injuries,fractures,osteoarthritis,patellofemoral joint pain

SUMMARY:
The aim of the study is to investigate Turkish validity and reliability of Marx Activity Rating Scale for patients with knee disorders.

DETAILED DESCRIPTION:
The aim of the study is to investigate Turkish validity and reliability of Marx Activity Rating Scale for patients with knee disorders.The study will include 30 patients with different types of knee disorders such as traumatic meniscal and ligament injuries,fractures,osteoarthtiris and patellofemoral joint pain.This study will conduct at Palmer&Still Physiotherapy Clinic.The original English form will be translated into Turkish according to guidelines.Subjects will complete translated Marx Activity Rating Scale,International Knee Documentation Committee (IKDC) subjective knee form and EuroQol EQ5D.Re-testing will be obtained after 1 month.

ELIGIBILITY:
Inclusion Criteria:

Older than 18 years can read and write Turkish have knee disorders such as traumatic mensical and ligament injuries,fractures,patellofemoral pain syndrome and/or mild osteoarthritis

Exclusion Criteria:

Individuals with multiple ligament injuries, large osteochondral fractures, large focal cartilage defects requiring surgery, malignancy, and advanced osteoarthritis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who have knee disorders such as traumatic mensical and ligament injuries,fractures,patellofemoral pain syndrome and/or mild osteoarthritis.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Marx Activity Rating Scale (MARS) | 1 month
  Knee-specific patient-reported outcome measure assesses the frequency of participation in sports-related activities for an adult population. It has a 5-point scale referring to the frequency of performing these activities in the past year.
  The maximum score is 16, while the minimum score is 0 for the patient. A higher score means more frequent sports-related participation.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Tuğçe Çil, Study Director — Yeditepe University
Locations (1):
- Palmer and Still Physiotherapy Clinic, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No